CLINICAL TRIAL: NCT05252533
Title: Open-label Study to Evaluate the Pharmacokinetics, Safety, and Immunogenicity of Ustekinumab in Pediatric Participants
Brief Title: A Study of Ustekinumab in Pediatric Participants (U-POPS) With Juvenile Psoriatic Arthritis or Psoriasis
Acronym: U-POPS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CR109159; CNTO1275ISD1001 (Other: Janssen Research and development, LLC)
Record Dates: First submitted 2022-02-16; First posted 2022-02-23 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Juvenile Psoriatic Arthritis; Psoriasis; Arthritis, Juvenile
MeSH Terms: conditions — Arthritis, Juvenile; Psoriasis | interventions — Ustekinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Juvenile Psoriatic Arthritis (jPsA) (Experimental): Participants (aged greater than or equal to [>=] 5 to less than [<] 18 years) will receive ustekinumab at the dose and frequency as prescribed by their treating health care professional (HCP).
  Interventions: Drug: Ustekinumab
- Cohort 2: Pediatric Psoriasis (PsO) (Experimental): Participants (aged >=6 to <18 years) will receive ustekinumab at the dose and frequency as prescribed by their treating HCP.
  Interventions: Drug: Ustekinumab

INTERVENTIONS:
Drug: Ustekinumab — This study does not provide dosing instructions for ustekinumab but will engage participants who have been treated with ustekinumab by their corresponding HCPs independent of this study.
  Other Names: STELARA

SUMMARY:
The purpose of the study is to evaluate pharmacokinetics (PK) of ustekinumab in juvenile psoriatic arthritis (jPsA) and pediatric psoriasis (PsO).

DETAILED DESCRIPTION:
jPsA is a complex, chronic, progressive, debilitating musculoskeletal disease with significant remaining medical need. There is a need for medications which have a similar efficacy profile and a well-characterized safety profile relative to currently available tumor necrosis factor alpha (TNF alpha) inhibitors for jPsA participants with active disease. STELARA (ustekinumab) is a fully human immunoglobulin G1 kappa monoclonal antibody which binds with high affinity to the p40 subunit common to both interleukin (IL)-12 and IL 23 preventing IL-12/23p40 binding to the IL 12 Rb1 cell surface receptor shared by both cytokines. Through this mechanism of action, ustekinumab effectively neutralizes IL-12 T helper 1- and IL-23 T helper 17-mediated cellular responses. Ustekinumab has been extensively studied in adult participants with psoriasis, psoriatic arthritis (PsA), Crohn's disease, and ulcerative colitis (UC). Additionally, ustekinumab has been studied in children (greater than or equal to [>=] 6 to less than [<] 12 years of age) and adolescents (>=12 to <18 years of age) with pediatric psoriasis [PsO]. This study consists of 3 visits: screening (Visit 1), interim and final visit (Visits 2 and 3) (Visits should be >=7 days apart). Key safety assessments include analyses of the incidence and types of adverse events (AEs), serious adverse events (SAEs), reasonably related AEs, and discontinuation of ustekinumab due to an AE, infections, and/or injection site and hypersensitivity reactions. Any newly identified malignancy, case of active tuberculosis (TB), or opportunistic infection will also be assessed. The total duration of the study is up to 20 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to (>=) 5 to less than (<) 18 years of age, inclusive, with a diagnosis of juvenile psoriatic arthritis (jPsA) (that is, International League Against Rheumatism [ILAR] or Vancouver criteria) by qualified health care professional (HCP)
* >=6 to <18 years of age, inclusive, with a diagnosis of pediatric psoriasis (PsO) by a qualified HCP
* Initiated ustekinumab treatment >=16 weeks prior to enrollment and received 3 or more doses of ustekinumab prior to enrollment
* Parent(s) (preferably both if available or as per local requirements) (or their legally acceptable representative) must sign an informed consent form (ICF) indicating that he or she understands the purpose of, and procedures required for, the study and is willing to allow the child to participate in the study. Assent is also required of children capable of understanding the nature of the study (typically 7 years of age and older) as described in informed consent process

Exclusion Criteria:

* Has poor tolerability of venipuncture or lack of adequate venous access for required blood sampling
* Has any condition that, in the opinion of the investigator, participation would not be in the best interest of the participant (example, compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments
* If currently enrolled in an investigational study, contact the study responsible physician to discuss eligibility for inclusion in study

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2022-05-24 (Actual); Primary Completion 2024-01-26 (Actual); Study Completion 2024-01-26 (Actual)

PRIMARY OUTCOMES:
Serum Concentration of Ustekinumab | Up to 16 weeks
  Serum samples will be analyzed to determine concentrations of ustekinumab using a validated, specific, and sensitive immunoassay method.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Up to 20 weeks
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Number of Participants with Serious Adverse Events (SAEs) | Up to 20 weeks
  An SAE is any untoward medical occurrence that at any dose: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; is a suspected transmission of any infectious agent via a medicinal product; is medically important.
Number of Participants with Antibodies to Ustekinumab | Up to 16 weeks
  Number of participants with antibodies to ustekinumab will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (10):
- United States (10):
  - Newport Huntington Medical Group, Huntington Beach, California
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Northwestern University Feinberg School of Medicine Ann & Robert H Lurie Children's Hospital, Chicago, Illinois
  - Michigan Dermatology Institute, Waterford, Michigan
  - Columbia University Medical Center, New York, New York
  - Akron Children s Hospital, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Pediatric Rheumatology Consultants of Austin, Austin, Texas

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Lam E, Berezny K, Bishop CJ, Lomax KG, Liva SG, Brunner HI, Paller AS, Diaz LZ, Lee LW, Rubin C, Carrasco R, Imundo L, Majlessi A, Smith V, Zhang R, Leu JH; U-POPS Study Group. Pharmacokinetics and Safety of Ustekinumab in Patients with Juvenile Psoriatic Arthritis: Results of the Real-World Ustekinumab Pediatric Opportunistic Pharmacokinetics Study (U-POPS). Rheumatol Ther. 2026 Feb;13(1):265-278. doi: 10.1007/s40744-025-00820-3. Epub 2025 Dec 26. PMID 41452420